CLINICAL TRIAL: NCT01983254
Title: Improving Psychological Distress Among Critical Illness Survivors and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); University of Pittsburgh (Other); University of Washington (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00043171; PCORI PFA 195 (Other Grant/Funding Number: PCORI PFA 195)
Record Dates: First submitted 2013-11-01; First posted 2013-11-13 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Intensive Care Unit Survivors; Informal Caregivers (Family and Friends)
Keywords: coping; acute respiratory failure; critical illness; depression; anxiety; post-traumatic stress; intensive care unit
MeSH Terms: conditions — Critical Illness; Depression; Anxiety Disorders | interventions — Early Intervention, Educational

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coping skills training (Experimental): 6 sessions of weekly telephone-based coping skills training delivered by trained interventionist
  Interventions: Behavioral: coping skills training
- education program (Active Comparator): 6 week access to a web-based, critical illness-specific education program
  Interventions: Other: education program

INTERVENTIONS:
Behavioral: coping skills training — 6-session coping skills training program delivered by telephone w/ web augmentation
  Arms: Coping skills training
Other: education program — web-based, ICU-specific education program
  Arms: education program

SUMMARY:
Patients who receive life support in intensive care units commonly suffer from persistent depression, anxiety, and post-traumatic stress disorder (PTSD) symptoms after discharge. We are trying to learn which is a better way to manage this distress: a telephone-based adaptive coping skills training program or an educational program.

DETAILED DESCRIPTION:
Public Summary of Research Project Why is this important? Nearly 800,000 Americans receive mechanical ventilation for acute respiratory failure in the ICU each year. Afterward, over half of both patients and their family caregivers suffer from psychological distress (depression, anxiety, and post-traumatic stress ["PTSD"]) for over 1 year after discharge. Patients and families told us that they need help with their distress because it worsens their quality of life. More specifically, patients said that learning how to adapt (that is, how to cope) with the physical and emotional changes of critical illness would be helpful. In fact, most ICU survivors use coping skills infrequently, which worsens psychological distress. But patients also told us that they wanted more information about critical illness, recovery, and what to expect. A lack of information increases PTSD symptoms. However, there are few treatments for this distress that can overcome ICU survivors' physical disability, great distance from expert medical centers, and concerns about how much treatments would cost. Therefore, we developed two treatments to address coping and lack of information.

What is the main goal? We aim to compare which of two treatments are more effective in reducing psychological distress and improving quality of life. One is a coping skills training (CST) program provided by telephone. The other is an education program about critical illness that is accessed primarily online. Also, we will determine if unique groups of people with special characteristics have especially good improvement-and if so, what personal factors explain this response.

How will we know which treatment is better? We will determine which treatment is most helpful by comparing participants' levels of psychological distress and quality of life with surveys taken over 6 months. We'll also record patients' own descriptions of how the treatments impacted their daily lives. The study will take 3 years and would be performed at 5 medical centers across the US that treat patients with diverse backgrounds and illnesses. 200 ICU survivor-family member pairs will be randomly assigned (like a coin flip) to receive either the CST program or the education program. Treatments consist of 6 weekly telephone calls with a trained staff member, web-based modules, and handouts.

How will this help others in the future? This research is important because it aims to improve long-term recovery for entire families by focusing on a devastating, common, yet inadequately addressed problem. These treatments were developed with the direct input of patients and families. These treatments represent a new direction in treating critical illness because they can be delivered inexpensively by phone, easily adapted to future technologies, overcome barriers to care common to ICU survivors, and shared easily by phone or computer with others in need across the world.

ELIGIBILITY:
Patient inclusion criteria:

* age >=18 and
* mechanical ventilation for more than 48 consecutive hours

Patient exclusions (pre-consent):

* current significant cognitive impairment (>=3 errors on the Callahan scale) or lacks decisional capacity
* pre-existing significant cognitive impairment
* residence at location other than home before hospital admission
* need for a translator because of poor English fluency [many study instruments are not validated in other languages]
* expected survival <3 months
* discharged to hospice (outpatient or inpatient)
* not liberated from mechanical ventilation at discharge

Additional patient exclusion criteria (present post-consent but pre-randomization):

* Patients will become ineligible if they become too ill to participate
* they develop significant cognitive disability, exhibit suicidality, they do not return home within 2 months after hospital discharge, or die.

Informal caregiver inclusion criteria:

* age >=18 years
* person most likely to provide the most post-discharge care.

Exclusions for caregivers are:

* history of significant cognitive impairment
* English fluency poor enough to require a medical translator

Informal caregiver exclusion criteria present after consent but before randomization:

* no longer available
* become too ill to participate
* exhibit suicidality

A total of 200 patient-caregiver dyads (total cohort = 400) are targeted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Cox, MD MPH, Principal Investigator — Duke University
Locations (4):
- United States (4):
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Cox CE, Porter LS, Hough CL, White DB, Kahn JM, Carson SS, Tulsky JA, Keefe FJ. Development and preliminary evaluation of a telephone-based coping skills training intervention for survivors of acute lung injury and their informal caregivers. Intensive Care Med. 2012 Aug;38(8):1289-97. doi: 10.1007/s00134-012-2567-3. Epub 2012 Apr 18. PMID 22527082
- [Result] Cox CE, Hough CL, Carson SS, White DB, Kahn JM, Olsen MK, Jones DM, Somers TJ, Kelleher SA, Porter LS. Effects of a Telephone- and Web-based Coping Skills Training Program Compared with an Education Program for Survivors of Critical Illness and Their Family Members. A Randomized Clinical Trial. Am J Respir Crit Care Med. 2018 Jan 1;197(1):66-78. doi: 10.1164/rccm.201704-0720OC. PMID 28872898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 417 participants were enrolled (277 patients and 140 informal caregivers). 261 participants were randomized (175 patients and 86 caregivers).
Period: Overall Study
Arm/Group | Coping Skills Training | Education Program
Started | 125 (86 patients, 39 caregivers) | 136 (89 patients, 47 caregivers)
Interview 1 | 125 (86 patients, 39 caregivers) | 136 (89 patients, 47 caregivers)
Interview 2 | 95 (65 patients, 30 caregivers) | 110 (71 patients, 39 caregivers)
Interview 3 | 91 (62 patients, 29 caregivers) | 106 (69 patients, 37 caregivers)
Completed | 91 (62 patients, 29 caregivers) | 106 (69 patients, 37 caregivers)
Not Completed | 34 | 30
Not completed — Death | 6 | 6
Not completed — Lost to Follow-up | 17 | 16
Not completed — too ill | 11 | 8

BASELINE CHARACTERISTICS:
Population: This includes 86 patients and 39 caregivers (coping skills training group) plus 89 patients and 47 caregivers (education program group).
Groups:
- Total: Total of all reporting groups
Arm/Group | Coping Skills Training | Education Program | Total
Number analyzed (Participants) | 125 | 136 | 261
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 105 | 110 | 215
  >=65 years | 20 | 26 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Separate tables are shown for patients (n=175) and family members (n=86).
  years
    Patients: number analyzed (Participants) | 86 | 89 | 175
    Patients | 49.7 (13.8) | 53.7 (13.5) | 51.7 (13.8)
    Caregivers: number analyzed (Participants) | 39 | 47 | 86
    Caregivers | 50.0 (14.9) | 52.9 (15.2) | 51.4 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 73 | 144
  Male | 54 | 63 | 117
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 125 | 133 | 258
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 25 | 25 | 50
  White | 95 | 102 | 197
  More than one race | 1 | 5 | 6
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 125 | 136 | 261

OUTCOME MEASURES:

1. Primary Outcome: Hospital Anxiety and Depression Scale Score
Description: Hospital Anxiety and Depression Scale (HADS) questionnaire: The HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression. The anxiety and depression subscales each range from 0 to 21, with higher scores indicating higher anxiety/depression complains. Patients were defined as having anxiety or depression or both if the score was 8 or more in the corresponding subscale. The 3 month measure is primary outcome timing, though changes at 6 months will be tested as well
Time Frame: 3 & 6 months post-randomization
Population: Patients who completed the HADS scale at 3 & 6 months post-randomization.
Measure: Mean (Standard Error); unit: units on a scale (HADS summary score)
Arm/Group | Coping Skills Training | Education Program
Number analyzed (Participants) | 65 | 71
units on a scale (HADS summary score)
  3 months | 16.6 (0.9) | 15.3 (0.9)
  6 months: number analyzed (Participants) | 62 | 69
  6 months | 15.6 (1.0) | 15.9 (1.0)

2. Secondary Outcome: Impact of Events Scale-revised (IES-R) Score
Description: The IES-R evaluates subjective distress caused by traumatic events and assesses manifestations of post-traumatic stress disorder (PTSD) or acute stress disorder. It is not diagnostic but possesses excellent reliability and validity for manifestations of PTSD. The IES-R has three subscales (eight items on intrusion, eight items on avoidance, and six items on hyperarousal). Each item is scored on a four point scale: 0 = "not at all," 1 = "a little bit," 2 = "moderately often," 3 = "quite a bit," and 4 = "extremely often." The total score of each subscale may be averaged and a cumulative score of 30 is indicative of the presence of PTSD. The maximum score for each subscale is 32 for intrusion, 32 for avoidance, and 24 for hyperarousal. The minimum cumulative score is 0 and the maximum cumulative score possible is 88.3 months post-randomization is main time point while The 3 month IES-R score will be the primary analysis, though 6 month changes will be tested as well.
Time Frame: 3 & 6 months post-randomization
Population: Patients who completed the IES-R scale at 3 & 6 months post-randomization.
Measure: Mean (Standard Error); unit: units on a scale (IES-R)
Arm/Group | Coping Skills Training | Education Program
Number analyzed (Participants) | 65 | 71
units on a scale (IES-R)
  3 months | 31.0 (2.6) | 27.9 (2.6)
  6 months: number analyzed (Participants) | 62 | 69
  6 months | 29.4 (2.9) | 25.8 (2.9)

3. Other Pre Specified Outcome: Total Weeks at Home Post-randomization
Description: here reported as weeks (instead of days) not at home for simplicity
Time Frame: over 6 months follow up
Population: patients
Measure: Mean (Standard Deviation); unit: weeks not at home during follow up
Units Other Than Participants: weeks
Arm/Group | Coping Skills Training | Education Program
Number analyzed (Participants) | 69 | 75
Number analyzed (weeks) | 24 | 24
weeks not at home during follow up | 1.3 (3.0) | 1.6 (3.5)

ADVERSE EVENTS:
Arm/Group | Coping Skills Training | Education Program
All-Cause Mortality (participants affected / at risk) | 6/125 | 6/136
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/136
Other Adverse Events (participants affected / at risk) | 0/125 | 0/136

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No